CLINICAL TRIAL: NCT03044639
Title: Four Parenteral Lipid Emulsions and the Liver Function
Brief Title: Parenteral Lipid Emulsions and the Liver Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanley Dudrick's Memorial Hospital (Other)
Responsible Party: Principal Investigator, Stanislaw Klek, Head of the Department, Stanley Dudrick's Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IVLE
Record Dates: First submitted 2017-01-22; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-01

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure | interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, multi-centric study performed in four parallel groups
Who Masked: Investigator
Masking Description: No information on the lipid emulsion's type provided neither to the patient nor the leading physician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Provision of LCT emulsions in PN (Experimental): Intervention: Lipid Emulsions, Intravenous. Daily provision of LCT-based lipid emulsion as a part of parenteral nutrition along with dextrose, amino acids, electrolytes, trace elements, vitamins and water in the dose of 0.8-1.0 g/kg/day.
  Interventions: Drug: Lipid Emulsions, Intravenous
- Provision of MCT/LCT emulsions in PN (Experimental): Intervention: Lipid Emulsions, Intravenous. Daily provision of MCT/LCT lipid emulsion as a part of parenteral nutrition along with dextrose, amino acids, electrolytes, trace elements, vitamins and water in the dose of 0.8-1.0 g/kg/day.
  Interventions: Drug: Lipid Emulsions, Intravenous
- Provision of Olive oil emulsions in PN (Experimental): Intervention: Lipid Emulsions, Intravenous. Daily provision of Olive-oil/ LCT lipid emulsion as a part of parenteral nutrition along with dextrose, amino acids, electrolytes, trace elements, vitamins and water in the dose of 0.8-1.0 g/kg/day.
  Interventions: Drug: Lipid Emulsions, Intravenous
- Provision of SMOF lipid emulsions in PN (Experimental): Intervention: Lipid Emulsions, Intravenous. Daily provision of SMOF lipid emulsion as a part of parenteral nutrition along with dextrose, amino acids, electrolytes, trace elements, vitamins and water in the dose of 0.8-1.0 g/kg/day.
  Interventions: Drug: Lipid Emulsions, Intravenous

INTERVENTIONS:
Drug: Lipid Emulsions, Intravenous — The every day provision of lipid emulsion as a part of parenteral nutrition along with dextrose, amino acids, electrolytes, trace elements, vitamins and water in the dose of 0.8-1.0 g/kg/day.
  Other Names: parenteral lipid provision

SUMMARY:
The randomized, double-blind, multi-centric study performed in four parallel groups to compare all lipid emulsions, which can be used as a part of PN. Patients with home parenteral nutrition due to stable intestinal failure, were randomly assigned to receive parenteral nutrition with one the following lipid emulsions:

* Long-chained triglycerides (LCT group)
* Medium/ long-chained triglycerides MCT/LCT (50:50, MCT/LCT group))
* Olive oil/ LCT (80:20, OO group))
* SMOFlipid (Omega-3/ olive oil/ MCT/ LCT, SMOF group)

DETAILED DESCRIPTION:
Intravenous lipid emulsion (IVLE) is the essential component of parenteral nutrition (PN), because it is a very efficient source of energy and essential fatty acids (FA).The prevalence of abnormal liver function tests during PN varies from 15 to 85%, according to most authors.[19-21] The severity of IFALD depends also on underlying disease, especially ongoing sepsis and pre-existing liver disease. A study comparing all lipid emulsions, which can be used as a part of PN, has never been done. The aim of the study was to compare the clinical value of the four most popular intravenous lipid emulsions in regards to the liver function in long term intestinal failure patients.Patients with home parenteral nutrition due to stable intestinal failure, were randomly assigned to receive parenteral nutrition with one the following lipid emulsions:

* Long-chained triglycerides (LCT group)
* Medium/ long-chained triglycerides MCT/LCT (50:50, MCT/LCT group))
* Olive oil/ LCT (80:20, OO group))
* SMOFlipid (Omega-3/ olive oil/ MCT/ LCT, SMOF group) Randomization was performed after assessment and check for in-/exclusion criteria if the patient has met all study eligibility requirements.

The test emulsion became a part of regular PN admixture, which was used to feed patient at home. The study was performed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. chronic intestinal failure (CIF) receiving HPN including lipids
2. metabolic stability on HPN for more than three months (metabolic stability = the absence of pathological laboratory resulting in the change of PN regime for at least one month)
3. 1.0 g lipids/kg body weight per day as a part of PN

Exclusion Criteria:

1. Existing liver failure: an elevation of SGOT, SGTP, total bilirubin, GGTP, alkaline phosphatase of more than 1.5 times x normal value
2. Patients in whom PN was interrupted for longer than 4 continuous weeks in the preceding 6 months
3. Patients with history of cancer and anti-cancer treatment within the last 5 years
4. Severe hyperlipidemia
5. Severe coagulopathy
6. Severe renal insufficiency
7. Acute thromboembolic events
8. Positive test for HIV, Hepatitis B or C (from medical history)
9. Known or suspected drug or alcohol abuse
10. Participation in another interventional clinical trial in parallel or within three months prior to the start of this clinical trial
11. For women with childbearing potential (i.e. females who are not chemically or surgically sterile or females who are not postmenopausal) or women of childbearing potential tested positive on standard pregnancy test (urine dipstick) or/ and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-04-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Liver function | 12 months
  Measurement of bilirubin - at the beginning and every three months up to 12 months

SECONDARY OUTCOMES:
Liver function 2 | 12 months
  Measurement of SGTP - at the beginning and every three months up to 12 months
Liver function 3 | 12 months
  Measurement of SGOT - at the beginning and every three months up to 12 months
Liver function 4 | 12 months
  Measurement of GGTP - at the beginning and every three months up to 12 months
Liver function 5 | 12 months
  Measurement of alkaline phosphatase - at the beginning and every three months up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw Klek, MD PhD, Principal Investigator — Stanley Dudrick's Memorial Hospital
Locations (1):
- Stanley Dudrick's Memorial Hospital, Skawina, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calder PC. Hot topics in parenteral nutrition. Rationale for using new lipid emulsions in parenteral nutrition and a review of the trials performed in adults. Proc Nutr Soc. 2009 Aug;68(3):252-60. doi: 10.1017/S0029665109001268. Epub 2009 May 11. PMID 19426581
- [Background] Calder PC, Jensen GL, Koletzko BV, Singer P, Wanten GJ. Lipid emulsions in parenteral nutrition of intensive care patients: current thinking and future directions. Intensive Care Med. 2010 May;36(5):735-49. doi: 10.1007/s00134-009-1744-5. Epub 2010 Jan 14. PMID 20072779
- [Derived] Klek S, Szczepanek K, Scislo L, Walewska E, Pietka M, Pisarska M, Pedziwiatr M. Intravenous lipid emulsions and liver function in adult chronic intestinal failure patients: results from a randomized clinical trial. Nutrition. 2018 Nov;55-56:45-50. doi: 10.1016/j.nut.2018.03.008. Epub 2018 Mar 22. PMID 29960156